CLINICAL TRIAL: NCT04901793
Title: Efficacy of Virtual Reality in Pain Reduction in Orthopedic Pediatric Patients Measured by Patient Feedback and Heart Rate Monitoring
Brief Title: Efficacy of Virtual Reality in Pain Reduction in Orthopedic Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Lawrence Haber, Principal Investigator, Ochsner Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017.522
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2019-06

CONDITIONS: Orthopedic Disorder; Fractures, Bone
MeSH Terms: conditions — Musculoskeletal Diseases; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: A non-blinded computer-randomized prospective trial with two parallel study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Intervention Group (Experimental): Patient is fitted with a Virtual Reality headset and handheld remote control. Subject is able to play an interactive game during the duration of the in-office procedure.
  Interventions: Behavioral: Virtual Reality Headset and handheld remote control.
- Control Group (No Intervention): standard of care

INTERVENTIONS:
Behavioral: Virtual Reality Headset and handheld remote control. — Brand name: Oculus Quest
  Arms: Virtual Reality Intervention Group

SUMMARY:
To prospectively determine if pediatric patients undergoing orthopedic procedures can benefit from employing virtual reality for pain management.

DETAILED DESCRIPTION:
INTRODUCTION

Pediatric patients are exposed to procedures that can result in pain and anxiety. The International Association Study of Pain 2011 defines pain as an unpleasant sensory and emotional experience associated with actual or potential tissue damage. Pharmacological interventions have been used but consequences of this therapy, specifically opioids, are of concern. Distraction techniques have been implemented recently but there is a significant range of these techniques such as breathing, music, and play therapy, among others.

Some studies indicate child preferences and temperament can optimize outcomes in regards to therapy. Non-pharmacological analgesics have been shown to benefit patients overall. Watching videos, biofeedback, mental imagery, and hypnosis have all been reported to have analgesic effects in the literature. Additionally cognitive behavioral strategies particularly distraction have been shown to reduce pain reports as high as 85% of patients. The most recent emerging technique is virtual reality.

Virtual reality creates the illusion that user is immersed in another environment. A three dimensional world is seen through the eyepieces, and the user can interact with the world in several ways: by moving their head and neck to look around the environment and a hand held trigger allows you to shoot at objects within the environment. Because this is a more interactive environment and more attention capturing than simple distractions, VR is thought to be more beneficial than basic distraction techniques. Additionally, using a head-mounted display (HMD) prevents visual perception of the real world, decreasing the chance of distraction. Previous uses of distraction show that children only pay attention to the distraction for 2/3 of the procedure, but virtual reality prevents the distraction of the procedure's visual stimuli.

In this study the investigators will attempt to determine the benefit of using virtual reality distraction techniques with a head-mounted display in standard orthopedic consultations that involve pain. The literature review indicates that excepting burns, this study has not been performed previously. Additionally heart rate monitoring has not been previously been included in the analysis of pain reduction. The investigators will assess pain reduction using patient feedback and pain scales, but also heart rate monitoring pre-procedure, during procedure, and post-procedure. In this study, the only procedure will be cast removal.

OBJECTIVE

To prospectively determine if pediatric patients undergoing orthopedic procedures can benefit from employing virtual reality for pain management.

SPECIFIC AIMS

To identify any benefits from virtual reality use as pain management in the pediatric population by means of patient feedback and by heart rate monitoring during orthopedic care. By doing this we can determine if virtual reality should become a standard of care in pain management for the pediatric population.

RATIONALE AND SIGNIFICANCE Post-surgical pain has been reported to be difficult to manage and can potentially limit outcomes in the pediatric population. Pharmacologic management is not ideal and intolerable for some patients. In 2009, a study of 182 children in the burns and orthopedic department at Royal Children's Hospital, Brisbane, Australia, found that multimodal distraction devices (MMD) reduced pain and anxiety significantly as well as reduced future procedural pain. Multimodal devices are interactive devices that prepare the child for a procedure and uses developmentally appropriate distraction stories and games to alleviate the pain. Virtual reality provides an alternative method with high rewards.

In a case study of post-surgical twice-daily physiotherapy regimen, using a subjective pain scale, it was found to reduce pain by 41.2% compared to the control patients. Studies looking at IV placement with VR in children suggest satisfaction for children, parents, and nurses. That study suggested analyzing affective pain, anxiety, overall satisfaction, and pain intensity. A literature review from 2008-2013 also found that distraction techniques would be a simple and efficient non-pharmacological acute pain relief strategy and should be implemented in pediatric care settings. It suggested further exploring the use of virtual reality, which was emerging at the time.

Virtual reality distraction has also been used in chemotherapy, during burn wound care, intravenous port access in pediatric patients, to reduce pain and anxiety for invasive medical procedures, to help adolescents with cerebral palsy endure physiotherapy, and to reduce preoperative anxiety. Another study of VR during routine blood draw, found that VR was more effective than the standard of care for reducing pain and anxiety. They determined VR has the capacity to act as a preventive intervention transforming the blood draw experience into a potentially pain-free routine medical procedure particularly for patients with high anxiety. VR has the potential to both reduce outcomes for children but also reduce distress in their caregivers.

Uncontrolled pain is thought to have serious psychological and physiological consequences, including an increased risk of morbidity and even mortality in children. Recent estimates have shown that around 27% of children experience moderate to severe pain in the hospital; teenagers and infants experience higher amounts of 38% and 32% respectively. Pediatric patients with untreated pain are more susceptible to developing sensitization, hyperalgesia, chronic pain, and allodynia. Long-term effects can include alterations in circuitry that impact pain processing in the future which predispose to decreased sensitivity or hypersensitivity to painful stimuli.

METHODS/PROCEDURE

Patients who present to have a cast removed, percutaneous bone pin removed, or cast applied will undergo heart rate monitoring via a pulse oximeter and give feedback post-procedure. Patients will be selected if they are between the ages of 5 and 18 years of age, have no significant co-morbidities, and are not undergoing an emergent procedure. Approximately 100 patients will be enrolled in the study, with 50 participants in each of two groups. The two groups will be the intervention group- those with the VR headset, and a control group- those without a VR headset. The groups will be randomized, and demographic data including age and sex will be obtained. Patients who qualify for the study will be consented by a member of the study team during the visit.

The two groups will be randomized via GraphPad software through https://www.graphpad.com/quickcalcs/randomize2/. The website will randomly assign 50 subjects each to two groups, for a total of 100 subjects. The results will be copied into a secure computer database to keep track of the assigned groups. Patients will be assigned a study number from 001 through 100, according to the chronological order in which they are consented. From there, the investigators will match up the patient's study number with the results from GraphPad and determine the patient's group assignment.

Enrolled patients will be located at the Ochsner Medical Center, New Orleans, Louisiana. There will be no charges to the patient and no reduction of patient care. If the patient requires admission for management of their pain, they will be admitted to the inpatient unit and followed by the team. Patients will undergo heart rate monitoring before, during, and after the cast removal procedure. All patient data collected will be de-identified and stored on a secured database.

We will analyze our data with T-tests with 2-tailed and 2-sample unequal variance as the parameters.

PROTOCOL

This study will involve patients in the pediatric orthopedic setting at Ochsner Medical Center in New Orleans, Louisiana. This will be a prospective consecutive case series to evaluate the severity and reduction of pain in the pediatric population.

Randomization of study groups will be performed prior to any patient enrollment. There will be two study groups with approximately 50 subjects in each group. Participants in group 'A' will be fitted with the VR headset during their procedure. Participants in group 'B' will not be fitted with the VR headset and they will act as the control group. Prior to enrollment in this study, all patients will be properly informed and consented about the requirements, risks, benefits, and other relevant information of the study.

Patients will experience the standard of care and any abnormalities or distress will be addressed. If the patients require admission for pain management, they will be admitted to Ochsner Medical Center. Patients will continue to be monitored for the utmost patient care. The anticipated number of participants in the study is about 100 patients.

All factors between the groups will be kept as similar as possible with any changes being formally documented. Patients will be given follow-up instructions that are consistent with the standard of care for cast removal. It is our goal to determine if virtual reality should become a standard of care in the pediatric population in regard to orthopedic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Presented for an in-office procedure after a primary orthopedic injury
* Willing to participate in the study.
* Between age of 5 and 18

Exclusion Criteria:

* Any condition limiting subject ability to perceive and communicate information including developmental delay, Cerebral Palsy, or Autism Spectrum Disorder.
* Limitations in subject ability to use the VR system including an inability to sit upright or bilateral upper extremity injuries

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate | Baseline HR measured 2 minutes pre-operation. Procedural HR measured during procedure.
  Change from baseline max HR to intra-procedural max HR

SECONDARY OUTCOMES:
Perceived Anxiety | measured within 5 minutes of procedure completion
  Visual Analog Scale (VAS) for perceived anxiety about the procedure
Perceived Pain | measured within 5 minutes of procedure completion
  Visual Analog Scale (VAS) for perceived pain during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sean Waldron, MD, Principal Investigator — Ochsner Health System; Lawrence Haber, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Health Center, Jefferson, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koller D, Goldman RD. Distraction techniques for children undergoing procedures: a critical review of pediatric research. J Pediatr Nurs. 2012 Dec;27(6):652-81. doi: 10.1016/j.pedn.2011.08.001. Epub 2011 Oct 13. PMID 21925588
- [Background] Steele E, Grimmer K, Thomas B, Mulley B, Fulton I, Hoffman H. Virtual reality as a pediatric pain modulation technique: a case study. Cyberpsychol Behav. 2003 Dec;6(6):633-8. doi: 10.1089/109493103322725405. PMID 14756928
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Li A, Montano Z, Chen VJ, Gold JI. Virtual reality and pain management: current trends and future directions. Pain Manag. 2011 Mar;1(2):147-157. doi: 10.2217/pmt.10.15. PMID 21779307
- [Background] Miller K, Rodger S, Bucolo S, Wang XQ, Kimble RM. [Multimodal distraction to relieve pain in children undergoing acute medical procedures]. Zhonghua Shao Shang Za Zhi. 2009 Oct;25(5):352-6. Chinese. PMID 19951557
- [Background] Gold JI, Mahrer NE. Is Virtual Reality Ready for Prime Time in the Medical Space? A Randomized Control Trial of Pediatric Virtual Reality for Acute Procedural Pain Management. J Pediatr Psychol. 2018 Apr 1;43(3):266-275. doi: 10.1093/jpepsy/jsx129. PMID 29053848